CLINICAL TRIAL: NCT02046434
Title: Phenylbutyrate Response As a Biomarker for Alpha-Synuclein Clearance From Brain
Brief Title: Phenylbutyrate Response as a Biomarker for Alpha-synuclein Clearance From the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-2808
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parkinson's Diesase (Experimental): Participant will take Glycerol Phenylbutyrate, participant has Parkinson's Disease
  Interventions: Drug: Glycerol Phenylbutyrate
- Control (Experimental): Participant does not have Parkinson's Disease, Participant will be taking glycerol phenylbutyrate
  Interventions: Drug: Glycerol Phenylbutyrate

INTERVENTIONS:
Drug: Glycerol Phenylbutyrate
  Other Names: Ravicti

SUMMARY:
This is a Phase I clinical trial of the FDA approved drug Glycerol Phenylbutyrate to see if phenylbutyrate can increase the removal of alpha-synuclein from the brain into the bloodstream. Alpha-synuclein forms abnormal protein deposits in dopamine neurons and is believed to cause the death of brain cells, leading to Parkinson's Disease.

DETAILED DESCRIPTION:
This is a Phase I clinical trial of phenylbutyrate in 20 Parkinson patients and 20 age- and sex-matched normal control subjects to see if phenylbutyrate can increase the removal of alpha-synuclein from the brain into the bloodstream. All subjects will receive 20 grams/day of phenylbutyrate in the liquid form phenylbutyrate-triglyceride taken as one teaspoonful three times per day with meals. Blood will be drawn on two days prior to starting phenylbutyrate to measure alpha-synuclein concentrations. Phenylbutyrate-triglyceride will then be started and the change in plasma alpha-synuclein will be measured on day 1, 7, 14, and 21 days while taking phenylbutyrate. After 21 days, the drug will be stopped and a final blood sample will be measured at 28 days to see if plasma alpha-synuclein has fallen to its pre-phenylbutyrate level. No effects on Parkinson symptoms are expected during this short trial. Please note that although taking any type of Parkinson's drugs for symptomatic treatment disqualifies you, if you and your neurologist are willing and able to have you off Parkinson medication for six weeks before and during the trial, you may be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease with mild symptoms;
* May be on treatment with dopamine agonists provided that the treating neurologist agrees:

  1. that the drugs can be stopped for at least three weeks prior to participating in the phenylbutyrate study, and
  2. for the 4-week duration of the study.
* Age and sex matched normal control subjects from spouses and the general population;
* In good general health;
* Controlled hypertension, or
* Controlled hypercholesterolemia with medication.

Exclusion Criteria:

* Pregnant women;
* Current treatment with:

  1. L-3,4-dihydroxyphenylalanine (L-DOPA);
  2. monoamine oxidase (MAO) inhibitors,
  3. catechol-O-methyl transferase (COMT) inhibitors;
  4. histone deacetylase (HDAC) inhibitors;
  5. prednisone or other corticosteroids, or
  6. probenecid.
* Severe cardiopulmonary disease such as:

  1. congestive heart failure, or
  2. emphysema requiring supplemental oxygen;
* Renal disease with serum creatinine greater than 2.5;
* History of:

  1. depression in the prior year;
  2. epilepsy;
  3. stroke;
  4. prior brain surgery;
  5. dementia, or
  6. psychosis.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Levels of alpha-synuclein in blood plasma | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Curt R Freed, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Center, Aurora, Colorado, United States

REFERENCES:
- [Derived] Wen ZQ, Lin J, Xie WQ, Shan YH, Zhen GH, Li YS. Insights into the underlying pathogenesis and therapeutic potential of endoplasmic reticulum stress in degenerative musculoskeletal diseases. Mil Med Res. 2023 Nov 9;10(1):54. doi: 10.1186/s40779-023-00485-5. PMID 37941072